CLINICAL TRIAL: NCT01024894
Title: A Phase I/IIa Dose Escalation Study in Asia of Repeated Administration of "CYT107" (Glyco-r-hIL-7) Added on Treatment in Genotype 1 HCV Infected Patients Resistant to Pegylated Interferon-alpha and Ribavirin
Brief Title: Dose Escalation Study of Interleukin-7 (IL-7) and Bitherapy in Asiatic HCV Patients Resistant to Bitherapy
Acronym: ECLIPSE 3
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-09
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: interleukin-7; immune-based therapies; hepatitis C; chronic hepatitis; resistance to Peg-interferon and ribavirin bitherapy; immune specific responses to HCV; taiwan; phase 1/2a; viral disease; liver disease
MeSH Terms: conditions — Hepatitis C; Hepatitis, Chronic; Virus Diseases; Liver Diseases | interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT107 (Experimental)
  Interventions: Drug: Interleukin-7

INTERVENTIONS:
Drug: Interleukin-7 — 3 dose levels: 3, 10 & 20 µg/kg. 4 administrations, 1 per week

SUMMARY:
This study is designed to evaluate the safety of biological active dose of a new experimental drug, IL-7, in combination with standard bi-therapy in Asiatic patients with Hepatitis C chronic infection identified as non responders to the standard bi-therapy alone.

DETAILED DESCRIPTION:
This is a Phase I/IIa inter-patient dose-escalation study assessing weekly doses of Interleukin-7 (CYT107) in Asiatic adult patients infected by virus of genotype 1 of Hepatitis C and resistant to standard treatment with Peg-Interferon and Ribavirin (bi-therapy).

The dose escalation is aimed at establishing the safety of a biologically active doses of CYT107 added to the combination therapy of pegylated interferon-alpha and ribavirin. At each dose level, study patients will receive one subcutaneous administration of CYT107 per week for a total of 4.

Groups of 3 to 6 patients will be entered at each dose level of CYT107. Three dose levels are planned.

Eligible patients initially receive bi-therapy for 6-10 weeks. Thereafter, CYT107 is added for a cycle of four weekly injections at a defined dose level while standard bi-therapy continues for 9 weeks after CYT107 treatment discontinuation. The patients are then followed on a regular basis until reaching 48 weeks after the CYT107 treatment. The duration of study is approximatively 60 weeks with 20-25 weeks of bi-therapy.

Participants will have 1 overnight hospitalization and 15 clinic visit on a period of 60 weeks.

During the visits the following may be done:

* medical history, physical examination, blood tests
* electrocardiograms (ECG)
* chest X-Ray
* liver/spleen imaging
* urine tests

ELIGIBILITY:
Main Inclusion Criteria:

* HCV Genotype 1 infected patients
* Absence of viral response to previous treatments with pegylated interferon-alpha plus ribavirin
* Metavir ≤ F3 assessed by biopsy in the last 12 months

Main Exclusion Criteria:

* Active infection by HBV
* Infection by HIV-1 and /or HIV-2
* Apart from HCV infection, presence of active infection requiring a specific treatment or a hospitalization
* Other liver disease
* Body mass index (BMI) > 30kg/m2
* Relapse after previous response to pegylated IFN alpha and ribavirin therapy
* Previous bi-therapy with pegylated IFN alpha and ribavirin not well tolerated (in particular treatment discontinuation)
* Any history of malignancy apart from curatively treated basal cell carcinoma or in situ cervical carcinoma
* History of clinical autoimmune disease or active auto-immune disease
* History of severe asthma, presently on chronic medications
* Significant cardiac or pulmonary disease
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
safety of biologically active doses of CYT107 added to a combination therapy by pegylated interferon-alpha and ribavirin in Asian patients with a chronic infection by a genotype 1 HCV not responding to this combination therapy | 12 weeks after start of CYT107

SECONDARY OUTCOMES:
Pharmacokinetics and pharmacodynamics of CYT107 in this patients population. | At short and mid terms follow-ups
potential anti-viral effect of CYT107 | 4 weeks and 12 weeks after start of CYT107
long-term safety and viral load variations | 24 and 48 weeks after the start of CYT107
immune specific response to HCV | 8 and 12 weeks after start of CYT107

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Long Chuang, MD, Study Chair — Kaohsiung Medical University
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chi Mei Medical Center, Tainan
  - Cathay General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taipei